CLINICAL TRIAL: NCT07216066
Title: First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of Intrathecally Administered ALN-SNCA in Participants With Early Parkinson's Disease
Brief Title: First-in-Human Study of ALN-SNCA in Adult Participants With Early Parkinson's Disease (PD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-SNCA-PD-2482; 2025-521431-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Parkinsons Disease
Keywords: Early Parkinsons disease; Motor and non-motor brain systems; Bradykinesia plus; Resting tremor; Rigidity; Postural instability; Cognitive impairment; Mood disorders; Sleep disturbances; Autonomic dysfunction
MeSH Terms: conditions — Parkinson Disease; Tremor; Muscle Rigidity; Cognitive Dysfunction; Mood Disorders; Parasomnias; Primary Dysautonomias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ALN-SNCA Dose Escalation (Experimental)
  Interventions: Drug: ALN-SNCA
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-SNCA — Administered per the protocol
  Arms: ALN-SNCA Dose Escalation
Drug: Placebo — Administered per the protocol
  Arms: Matching Placebo

SUMMARY:
This study is researching an experimental drug called ALN-SNCA (called "study drug"). The study is focused on people with early Parkinson's disease, a disorder of the nervous system that affects movement. Parkinson's disease is caused by a gradual loss of nerve cells in the brain, especially those due to the harmful build-up of a protein called α-synuclein.

The aim of the study is to see if the study drug is safe and tolerated well enough to continue testing it in future studies and what side effects may happen from taking the study drug.

The study is looking at several other research questions, including:

* Whether the study drug can lower the level of α-synuclein protein in the Cerebrospinal Fluid (also referred to as "CSF", the fluid that surrounds the brain and spinal cord)
* How much study drug is in the blood, urine, and CSF at different times
* Compatible research to better understand the study drug (ALN-SNCA) and Parkinson's disease, including (but not limited to), whether the study drug can slow down the progression of Parkinson's disease symptoms

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of Parkinson's disease according to the Movement Disorder Society (MDS) criteria, as assessed by the investigator, with bradykinesia plus at least one of the other cardinal signs of Parkinson's disease (resting tremor, rigidity), without any other known or suspected cause of Parkinsonism
2. A diagnosis of Parkinson's disease for 4 years or less at the screening visit
3. Participant must meet one of the following criteria:

   1. Currently not receiving any standard-of-care (SoC) therapy for Parkinson's disease, has not been on oral dopaminergic therapy (ie, levodopa, dopamine agonists, or Monoamine Oxidase B [MAO-B] inhibitors) prior to dosing, and is not anticipated to require SoC therapy for Parkinson's disease within approximately 6 months following dosing, or
   2. Has been on a stable regimen of oral dopaminergic therapy for at least 3 months prior to dosing and is not anticipated to require dose adjustments within approximately 6 months following dosing
4. BMI ≤35 kg/m^2 at time of screening visit

Key Exclusion Criteria:

1. Medical history indicating a Parkinsonian syndrome other than Parkinson's disease, as defined in the protocol
2. Clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease (excluding Parkinson's disease) that, as assessed by the investigator, may confound the results of the study or pose an additional risk to the participant during study participation
3. Medical history of brain or spinal disease/injury that would interfere with the Lumbar Puncture (LP) procedure or CSF circulation, as defined in the protocol
4. Any contraindications to undergo a brain Magnetic Resonance Imaging (MRI)
5. An established allergy or intolerance to lidocaine anesthetic, as defined in the protocol
6. History of intolerance to Intrathecal (IT) injection(s)
7. Current history of bleeding diatheses that would increase risk of bleeding upon LP
8. Has undergone gene therapy, cell therapy or surgical treatment, including deep brain stimulation, for Parkinson's disease

NOTE: Other Protocol-defined Inclusion/Exclusion Criteria Apply

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2029-06-07 (Estimated); Study Completion 2029-06-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Through Week 80
Severity of TEAEs | Through Week 80

SECONDARY OUTCOMES:
Concentration of alpha (a)-synuclein protein in CSF | Through Week 48
Change from baseline in concentration of a-synuclein protein in CSF | Through Week 48
Concentration of ALN-SNCA in plasma | Through Week 48
Concentration of major metabolites in plasma | Through Week 48
Concentration of ALN-SNCA in CSF | Through Week 48
Concentration of major metabolites in CSF | Through Week 48
Fraction [fc] of ALN-SNCA excreted in urine | Over 24 hours
Fc of major metabolites excreted in urine | Over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Center for Human Drug Research, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/